CLINICAL TRIAL: NCT04299893
Title: Effectiveness and Cost-effectiveness of Ozone Therapy in Patients With Pain Secondary to Chemotherapy-induced Peripheral Neuropathy. Randomized, Triple-blind Clinical Trial (O3NPIQ)
Brief Title: Ozone Therapy in Chemotherapy-induced Peripheral Neuropathy: RCT (O3NPIQ)
Acronym: O3NPIQ
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bernardino Clavo, MD, PhD (Other)
Collaborators: Servicio Canario de Salud (Other); Instituto de Salud Carlos III (Other Government); Red de Investigación en Servicios de Salud en Enfermedades Crónicas (Other); Fundación DISA, Spain (Unknown); Fundación Española del Dolor (FED) (Unknown)
Responsible Party: Sponsor-Investigator, Bernardino Clavo, MD, PhD, MD, PhD, Head of Research Unit, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-156-1; PI 19/00458 (Other Grant/Funding Number: Instituto de Salud Carlos III); 016/2019 (Other Grant/Funding Number: Fundación DISA); BF1-19-03 (Other Grant/Funding Number: Fundación Española del Dolor (FED)); 2019-000821-37 (EudraCT Number)
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Pain, Neuropathic; Pain Syndrome
Keywords: complementary and integrative medicine; cost-effectiveness ratio; chemotherapy-induced peripheral neuropathy; pain; ozone therapy; quality of life related to health; shared decision-making tool; randomized controlled trial
MeSH Terms: conditions — Neuralgia; Somatoform Disorders; Pain | interventions — Ozone; Oxygen

STUDY DESIGN:
Intervention Model Description: Standard treatment + ozone therapy (O3/O2) versus Standard treatment + oxygen (O2) as placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) Masking of: patients, Medical Oncologists (clinical assessment), investigators obtaining other parameters (quality of life, biochemical and clinical parameters, hyperspectral images), investigators for statistical analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ozone Group (Experimental): Drug: Ozone Ozone Group: Usual treatment + Ozone therapy (O3/O2) by rectal insufflation. O3/O2 concentration progressively increased from 10 to 30 μg/ml; 40 sessions in 16 weeks.
  Other Names: O3
  Interventions: Drug: Ozone
- Control Group (Placebo Comparator): Drug: Oxygen Control Group: Standard treatment + Oxygen (O2) by rectal insufflation. O3/O2 concentration = 0 μg/ml (only O2); 40 sessions in 16 weeks.
  Other Names: O2
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Ozone — Ozone Group: Standard treatment + Ozone therapy (O3/O2) by rectal insufflation. O3/O2 concentration progressively increased from 10 to 30 μg/ml; 40 sessions in 16 weeks.
  Other Names: O3
  Arms: Ozone Group
Drug: Oxygen — Control Group: Standard treatment + Oxygen (O2) by rectal insufflation. O3/O2 concentration = 0 μg/ml (only O2); 40 sessions in 16 weeks.
  Other Names: O2
  Arms: Control Group

SUMMARY:
The main objective of this clinical trial is to evaluate the effectiveness and cost-effectiveness of adding ozone therapy to the clinical management of patients with pain secondary to chemotherapy-induced peripheral neuropathy

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) decreases the quality of life of patients and can lead to a decrease and/or interruption of the chemotherapy treatment-limiting its effectiveness. The therapeutic measures for the CIPN are very limited in their number and efficacy.

Main Objectives: 1) To evaluate the clinical effect on the health-related quality of life (HRQOL) of adding ozone to the usual patient´s treatment with persistent pain because of CIPN. 2) Estimate the additional costs and evaluate the cost-effectiveness ratio.

Secondary Objectives: To evaluate the evolution of 3) oxidative stress and chronic inflammation through biochemical measurements; 4) anxiety and depression of patients; 5) the diagnostic and predictive value of hyperspectral imaging in the assessment of pain; 6) the acceptability of patients to a shared decision-making (SDM) tool.

METHODOLOGY: Randomized controlled trial (RCT) phase II-III, randomized, triple-blind; 42 patients with any kind of cancer treated with any kind of chemotherapy, with CIPN of grade > = 2 for > = 3 months.

TREATMENT: All patients will receive: usual treatment + 40 rectal insufflation sessions of O3/O2 in 16 weeks:

* Ozone-Arm (n = 21): concentration of O3/O2 increasing from 10 to 30 μg/ml.
* Control-placebo- Arm (n = 21): concentration of O3/O2 = 0 μg/ml.

Main Variables: At the end of treatment with O3/O2 the following variables will be analyzed: 1) "average pain" secondary to CIPN following the Brief Pain Inventory-Short Form (BPI-SF); 2) health-related quality of life (HRQOL) and utilities using EQ-5D-5L and SF-36 quality of life questionnaires; 3) Direct costs.

Secondary Variables: 3) biochemical parameters of oxidative stress and inflammation; 4) Hamilton scale for anxiety and depression; 5) hyperspectral images; 6) acceptability of patients to a shared decision-making (SDM) tool.

Assessments at weeks: 0 (baseline), 16 (end of O3/O2 insufflations, objective), and 28 (end of follow-up, control).

Length of treatment: 16 weeks.

Follow-up: 12 weeks after finishing O3/O2 insufflation.

Planned length of the clinical trial: 36 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults > = 18 years old.
* 2. Any kind of cancer in any stage, treated with any kind of chemotherapy, and life expectancy > = 6 months.
* 3. Clinical diagnosis of painful chemotherapy-induced peripheral neuropathy, toxicity Grade 2 or higher according to the Common Toxicity Criteria for Adverse Events (CTCAE) from the National Cancer Institute of EEUU, v.5.0, for > = 3 months and without the inclusion of new treatments for pain and/or neuropathy for > = 1 month.
* 4. "Average pain" > = 3/10 according to the Brief Pain Inventory-Short Form (BPI-SF) > = 3 months beyond chemotherapy completion.
* 5. Pregnant women cannot participate in the clinical trial.
* 6. Before enrollment, women of childbearing potential should obtain a negative result in the serum or urine pregnancy test at the screening visit and accept the use of appropriate contraceptive methods at least from the 14 days prior to the first ozone therapy session up to 14 days after the last one.
* 7. Patients who have signed and dated the study 's specific informed consent

Exclusion Criteria:

* 1. Age < 18 years old.
* 2. Pregnancy at the time of enrollment.
* 3. Women with childbearing potential who are unwilling to perform a pregnancy test and/or employ adequate contraception from the 14 days prior to the first ozone therapy session up to 14 days after the last one.
* 4. Clinical suspicion that peripheral neuropathy (compressive or diabetic neuropathy) in the same area prior to receiving neurotoxic chemotherapy.
* 5. Psychiatric illness or social situations that would limit compliance with study requirements.
* 6. Those who are unable to fill in the scales used to measure quality of life variables
* 7. Specific liver enzymes [Aspartate Aminotransferase (AST), and Alanine Aminotransferase (ALT) > 5 times the upper limit of normal
* 8. Increased creatinine > 3 times the upper limit of normal.
* 9. Hemodynamically or clinically unstable patients or uncontrolled severe illness.
* 10. Uncontrolled cancer disease.
* 11. Leptomeningeal carcinomatosis.
* 12. Life expectancy < 6 months
* 13. Contraindication or disability for rectal ozone administration or to attend scheduled treatments.
* 14. Known allergy to ozone.
* 15.Patients who do not meet all the inclusion criteria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in "Average pain" according to the Brief Pain Inventory-Short Form (BPI-SF) (at the end of ozone therapy) | 16 weeks
  Self-reported evaluation of 15 items to assess the severity of pain on daily functions in seven interference areas. From the 15 items, 11 items are scored from 0 ("No pain" or "Does not no interfere") to 10 ("Pain as bad as you can imagine" or "Completely interferes").
Direct Hospital Cost (at the end of ozone therapy) | 16 weeks
  The direct expenses incurred by the hospital in providing services (medication, tests, medical visits...) during the 16 weeks of ozone therapy (in euros).

SECONDARY OUTCOMES:
Change from Baseline in quality of life by the "5-level, 5-dimension EuroQol" (EQ-5D-5L) questionnaire (at the end of ozone therapy) | 16 weeks
  Self-reported evaluation of: a) 5 physical and emotional items scored in five levels, from 1 (best: I have no problem) to 5 (worst: I have extreme problem or I am unable to…) and b) additional self-assessment of health by a visual analogue scale (0 = worst health patient can imagine, 100 = best health patient can imagine)
Change from Baseline in quality of life by the "Short Form 36-item health survey" (SF-36v2) questionnaire (at the end of ozone therapy) | 16 weeks
  Self-reported evaluation of 36 items (0 = worst, 100 = best). Final accumulated total range from 0 (worst) to 100 (best)
Change from Baseline in Biochemical parameters of oxidative stress (at the end of ozone therapy) | 16 weeks
  Serum levels of superoxide dismutase, glutathione, glutathione peroxidase and free radicals
Change from Baseline in Biochemical parameters of inflammation (at the end of ozone therapy) | 16 weeks
  Serum levels of pro-inflammatory interleukins and TNFalpha
Change from Baseline in Hyperspectral image of painful area (at the end of ozone therapy) | 16 weeks
  Assessment of the percentage of reflectance for each wavelength
Change from Baseline in Levels of anxiety and depression according to the Hamilton scale (at the end of ozone therapy) | 16 weeks
  Clinician-administered depression assessment scale with 17 items pertaining to symptoms of depression experienced over the past week. Each item is scored from 0 (better, no alteration) to 2 (worse level of alteration) for items with three options, or from or from 0 (better, no alteration) to 4 (worse level of alteration) for items with five options. Overall score is from 0 (better, no anxiety/depression) to 52 (worse, very severe anxiety/depression).
Change from Baseline in Nerve conduction studies in the painful area (at the end of ozone therapy) | 16 weeks
  Assessment of nerve conduction velocity (in m/s)
Incidence of severe adverse events in accordance with the definition of the Council for International Organizations of Medical Sciences (at the end of ozone therapy) | 16 weeks
  Number of events that are fatal, life threatening, leading to or prolonging a stay in hospital, or resulting in severe disability
Change from Baseline in "Average pain" according to the Brief Pain Inventory-Short Form (BPI-SF) (at 12 weeks after the end of ozone therapy) | 28 weeks
  Self-reported evaluation of 15 items to assess the severity of pain on daily functions in seven interference areas. From the 15 items, 11 items are scored from 0 ("No pain" or "Does not no interfere") to 10 ("Pain as bad as you can imagine" or "Completely interferes")
Direct Hospital Cost (at 12 weeks after the end of ozone therapy) | 28 weeks
  The direct expenses incurred by the hospital in providing services (medication, tests, medical visits...) during the 16 weeks of ozone therapy (in euros)
Change from Baseline in quality of life by the "5-level, 5-dimension EuroQol" (EQ-5D-5L) questionnaire (at 12 weeks after the end of ozone therapy) | 28 weeks
  Self-reported evaluation of: a) 5 physical and emotional items scored in five levels, from 1 (best: I have no problem) to 5 (worst: I have extreme problem or I am unable to…) and b) additional self-assessment of health by a visual analogue scale (0 = worst health patient can imagine, 100 = best health patient can imagine)
Change from Baseline in quality of life by the "Short Form 36-item health survey" (SF-36v2) questionnaire (at 12 weeks after the end of ozone therapy) | 28 weeks
  Self-reported evaluation of 36 items (0 = worst, 100 = best). Final accumulated total range from 0 (worst) to 100 (best)
Change from Baseline in Biochemical parameters of oxidative stress (at 12 weeks after the end of ozone therapy) | 28 weeks
  Serum levels of superoxide dismutase, glutathione, glutathione peroxidase and free radicals
Change from Baseline in Biochemical parameters of inflammation (at 12 weeks after the end of ozone therapy) | 28 weeks
  Serum levels of pro-inflammatory interleukins and TNFalpha
Change from Baseline in Hyperspectral image of painful area (at 12 weeks after the end of ozone therapy) | 28 weeks
  Assessment of the percentage of reflectance for each wavelength
Change from Baseline in Levels of anxiety and depression according to the Hamilton scale (at 12 weeks after the end of ozone therapy) | 28 weeks
  Clinician-administered depression assessment scale with 17 items pertaining to symptoms of depression experienced over the past week. Each item is scored from 0 (better, no alteration) to 2 (worse level of alteration) for items with three options, or from or from 0 (better, no alteration) to 4 (worse level of alteration) for items with five options. Overall score is from 0 (better, no anxiety/depression) to 52 (worse, very severe anxiety/depression)
Change from Baseline in Nerve conduction studies in the painful area (at 12 weeks after the end of ozone therapy) | 28 weeks
  Assessment of nerve conduction velocity (in m/s)
Incidence of severe adverse events in accordance with the definition of the Council for International Organizations of Medical Sciences (at 12 weeks after the end of ozone therapy) | 28 weeks
  Number of events that are fatal, life threatening, leading to or prolonging a stay in hospital, or resulting in severe disability

CONTACTS AND LOCATIONS:
Overall Officials: Bernardino Clavo, MD, PhD, Study Chair — Dr. Negrín University Hospital, Las Palmas, Spain; Pedro G Serrano-Aguilar, MD, PhD, Study Director — Servicio de Evaluación. Servicio Canario de Salud. Spain; Delvys Rodríguez-Abreu, MD, Principal Investigator — Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas, Spain; Gustavo M Callico, Prof, PhD, Principal Investigator — Institute for Applied Microelectronics, University of Las Palmas de G. C., Spain; Francisco Rodríguez-Esparragón, BSc, PhD, Principal Investigator — Dr. Negrín University Hospital, Las Palmas, Spain; Bernardino Clavo, MD, PhD, Principal Investigator — Dr. Negrín University Hospital, Las Palmas, Spain
Locations (2):
- Spain (2):
  - Complejo Hospitalario Materno Insular, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith EM, Pang H, Cirrincione C, Fleishman S, Paskett ED, Ahles T, Bressler LR, Fadul CE, Knox C, Le-Lindqwister N, Gilman PB, Shapiro CL; Alliance for Clinical Trials in Oncology. Effect of duloxetine on pain, function, and quality of life among patients with chemotherapy-induced painful peripheral neuropathy: a randomized clinical trial. JAMA. 2013 Apr 3;309(13):1359-67. doi: 10.1001/jama.2013.2813. PMID 23549581
- [Background] Durand JP, Deplanque G, Montheil V, Gornet JM, Scotte F, Mir O, Cessot A, Coriat R, Raymond E, Mitry E, Herait P, Yataghene Y, Goldwasser F. Efficacy of venlafaxine for the prevention and relief of oxaliplatin-induced acute neurotoxicity: results of EFFOX, a randomized, double-blind, placebo-controlled phase III trial. Ann Oncol. 2012 Jan;23(1):200-205. doi: 10.1093/annonc/mdr045. Epub 2011 Mar 22. PMID 21427067
- [Background] Albers JW, Chaudhry V, Cavaletti G, Donehower RC. Interventions for preventing neuropathy caused by cisplatin and related compounds. Cochrane Database Syst Rev. 2014 Mar 31;2014(3):CD005228. doi: 10.1002/14651858.CD005228.pub4. PMID 24687190
- [Background] Hershman DL, Lacchetti C, Dworkin RH, Lavoie Smith EM, Bleeker J, Cavaletti G, Chauhan C, Gavin P, Lavino A, Lustberg MB, Paice J, Schneider B, Smith ML, Smith T, Terstriep S, Wagner-Johnston N, Bak K, Loprinzi CL; American Society of Clinical Oncology. Prevention and management of chemotherapy-induced peripheral neuropathy in survivors of adult cancers: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2014 Jun 20;32(18):1941-67. doi: 10.1200/JCO.2013.54.0914. Epub 2014 Apr 14. PMID 24733808
- [Background] Bocci V, Borrelli E, Travagli V, Zanardi I. The ozone paradox: ozone is a strong oxidant as well as a medical drug. Med Res Rev. 2009 Jul;29(4):646-82. doi: 10.1002/med.20150. PMID 19260079
- [Background] Bocci VA, Zanardi I, Travagli V. Ozone acting on human blood yields a hormetic dose-response relationship. J Transl Med. 2011 May 17;9:66. doi: 10.1186/1479-5876-9-66. PMID 21575276
- [Background] Bocci V, Valacchi G. Nrf2 activation as target to implement therapeutic treatments. Front Chem. 2015 Feb 2;3:4. doi: 10.3389/fchem.2015.00004. eCollection 2015. PMID 25699252
- [Background] Clavo B, Ceballos D, Gutierrez D, Rovira G, Suarez G, Lopez L, Pinar B, Cabezon A, Morales V, Oliva E, Fiuza D, Santana-Rodriguez N. Long-term control of refractory hemorrhagic radiation proctitis with ozone therapy. J Pain Symptom Manage. 2013 Jul;46(1):106-12. doi: 10.1016/j.jpainsymman.2012.06.017. Epub 2012 Oct 26. PMID 23102757
- [Background] Clavo B, Rodriguez-Esparragon F, Rodriguez-Abreu D, Martinez-Sanchez G, Llontop P, Aguiar-Bujanda D, Fernandez-Perez L, Santana-Rodriguez N. Modulation of Oxidative Stress by Ozone Therapy in the Prevention and Treatment of Chemotherapy-Induced Toxicity: Review and Prospects. Antioxidants (Basel). 2019 Nov 26;8(12):588. doi: 10.3390/antiox8120588. PMID 31779159
- [Background] Clavo B, Martinez-Sanchez G, Rodriguez-Esparragon F, Rodriguez-Abreu D, Galvan S, Aguiar-Bujanda D, Diaz-Garrido JA, Canas S, Torres-Mata LB, Fabelo H, Tellez T, Santana-Rodriguez N, Fernandez-Perez L, Marrero-Callico G. Modulation by Ozone Therapy of Oxidative Stress in Chemotherapy-Induced Peripheral Neuropathy: The Background for a Randomized Clinical Trial. Int J Mol Sci. 2021 Mar 10;22(6):2802. doi: 10.3390/ijms22062802. PMID 33802143
- [Background] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Ozone Therapy in Refractory Pelvic Pain Syndromes Secondary to Cancer Treatment: A New Approach Warranting Exploration. J Palliat Med. 2021 Jan;24(1):97-102. doi: 10.1089/jpm.2019.0597. Epub 2020 May 5. PMID 32379556
- [Background] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Long-Term Results with Adjuvant Ozone Therapy in the Management of Chronic Pelvic Pain Secondary to Cancer Treatment. Pain Med. 2021 Sep 8;22(9):2138-2141. doi: 10.1093/pm/pnaa459. No abstract available. PMID 33738491
- [Background] Clavo B, Rodriguez-Abreu D, Galvan S, Federico M, Martinez-Sanchez G, Ramallo-Farina Y, Antonelli C, Benitez G, Rey-Baltar D, Jorge IJ, Rodriguez-Esparragon F, Serrano-Aguilar P. Long-term improvement by ozone treatment in chronic pain secondary to chemotherapy-induced peripheral neuropathy: A preliminary report. Front Physiol. 2022 Aug 30;13:935269. doi: 10.3389/fphys.2022.935269. eCollection 2022. PMID 36111149